CLINICAL TRIAL: NCT07202702
Title: Modulation of Motor Learning Via tDCS in a Dexterous Video Game Task
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Zachary Riley, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26243
Record Dates: First submitted 2025-08-18; First posted 2025-10-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: experimental and control groups
Who Masked: Participant
Masking Description: The subjects should not know which group they are in with the SHAM protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- tDCS (Experimental): This group will receive 20 minutes of 1 mA tDCS stimulation to the motor cortex while playing the videogame.
  Interventions: Device: tDCS
- SHAM (Placebo Comparator): This group will receive 30 seconds of 1 mA tDCS stimulation to the motor cortex and then it will shut off, effectively serving as a control, while subjects play the videogame for 20 minutes
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Applying tDCS to determine if it facilitates learning of a video game task

SUMMARY:
The purpose of this study is to determine whether "transcranial direct current stimulation" (tDCS) is effective in enhancing learning of complex motor tasks of precision and accuracy that require the simultaneous coordination of both hands. The study will utilize a between-subjects, SHAM controlled design. Subjects will be randomly selected to receive either SHAM (n=26) or a-tDCS (n=26) stimulation and will be blinded to their condition throughout testing. Subjects will complete a total of two testing sessions, separated by ~24 hours. Both sessions will have the subject play the videogame "Guitar Hero", with a single song done for several trials as pre- and post-assessments. The first session will contain a 20-minute practice/stimulation block where subjects practice the guitar task while receiving either "active" or "inactive" stimulation of the motor cortex. The first session will last approximately 75 to 90 minutes whereas the second session will last approximately 15 to 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 and 45 years old (to avoid any changes in the developing brain, or with aging).
* Answer 'no' to questions 2 through 16 on the tDCS checklist as these factors can increase likelihood of adverse events with tDCS
* No neurological damage, disease, or dysfunction (nerve damage, chronic pain disorders, diabetic neuropathy) that affect the upper limbs.
* No significant acute or chronic medical, neurologic, or illness in the patient that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study

Exclusion Criteria:

* • Currently prescribed and taking stimulant medication (Adderall, Ritalin, Vyvanse, etc.)

  * Consumption of over-the-counter stimulants such as caffeine or nicotine (coffee, soda, supplements, energy drinks, tobacco products, or other nicotine containing products such as gum, vape pens, etc...) 12 hours prior to entering the lab on the day of testing as this can directly affect cortical excitability. If a subject takes any of these substances 12 hours prior to session 1 they will be asked to reschedule for a later date.
  * Have played a real stringed instrument in the last 12 months (e.g. guitar, bass, violin)
  * Have played the videogame "Guitar Hero" on a traditional guitar controller in the last 12 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in a video game | 1 year
  To determine whether a-tDCS influences motor skill acquisition of a dexterous video game task by measuring the outcome of videogame performance (number of notes played) with and without a-tDCS

SECONDARY OUTCOMES:
Retention and Learning | 1 Year
  Learning will be measured within-groups by examining retention, or the outcome of video game performance (number of notes played) between the first and second sessions

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Riley, Principal Investigator — Indiana University
Locations (1):
- National Institute for Fitness and Sport, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No